CLINICAL TRIAL: NCT07276308
Title: The Roles of Psychophysiological Stress and Cognitive Markers on Perceptual Responses During Low-volume High-intensity Interval Exercise in Overweight-to-obese Adults
Brief Title: Psychophysiological and Cognitive Responses to Low-Volume High-Intensity Interval Exercise in Overweight-to-Obese Adults
Acronym: PSYCOG-HIIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Ruohan Zhang, Principal Investigator (PhD Candidate), Universiti Sains Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: USM/JEPeM/22080549; FRGS/1/2022/SKK06/USM/03/5 (Other Grant/Funding Number: Universiti Sains Malaysia)
Record Dates: First submitted 2025-11-14; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Overweight and/or Obesity; Overweight and Obese Adults
Keywords: Exercise; Psychophysiological Stress; Cognitive traits; Affective Responses; High-Intensity Interval Exercise; Perceptual Responses
MeSH Terms: conditions — Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-Volume High-Intensity Interval Exercise (Lv-HIIE) (Experimental): Participants will perform a low-volume high-intensity interval exercise (Lv-HIIE) program consisting of 6-10 cycling intervals at 90% of maximal aerobic speed, interspersed with 75-second active recovery periods. The intervention will be conducted three times per week for 10 weeks under supervised laboratory conditions. Each session will include standardized warm-up and cool-down phases. The study aims to evaluate psychophysiological stress, cognitive markers, and perceptual responses across repeated exercise sessions in overweight-to-obese adults.
  Interventions: Behavioral: Low-Volume High-Intensity Interval Exercise (Lv-HIIE)

INTERVENTIONS:
Behavioral: Low-Volume High-Intensity Interval Exercise (Lv-HIIE) — The intervention consists of a supervised low-volume high-intensity interval exercise (Lv-HIIE) program performed on a cycle ergometer. Each session includes 6-10 intervals of 1 minute at 90% of maximal aerobic speed, interspersed with 75-second active recovery periods. Participants will train three times per week for 10 weeks under laboratory supervision. Each session begins with a standardized 5-minute warm-up and ends with a 5-minute cool-down. The program is designed to investigate changes in psychophysiological stress (ACTH, cortisol), cognitive markers (goal orientation, hardiness), and perceptual responses (affective valence, perceived exertion, enjoyment) across repeated exercise exposures in overweight-to-obese adults.
  Other Names: Lv-HIIE Training; Low-Volume HIIE; High-Intensity Interval Exercise Program

SUMMARY:
This study aims to explore how stress-related hormones and psychological traits influence people's feelings and perceptions during a short and intense form of exercise called low-volume high-intensity interval exercise (Lv-HIIE). Adults with overweight or obesity participated in a supervised 10-week cycling program consisting of repeated one-minute high-intensity efforts separated by short recovery periods.

The research examines how psychophysiological stress markers (such as cortisol and ACTH), cognitive traits (such as goal orientation and hardiness), and perceptual responses (such as exertion, mood, and enjoyment) change over time. Findings from this study may help develop exercise programs that are more enjoyable, sustainable, and personalized for individuals with higher body-mass categories.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between the ages of 20-35 years old
* BMI of 23 kg.m² to 30 kg.m2
* Medically fit to exercise.
* Physically inactive individuals (do not achieve 150 minutes of moderate-intensity exercise/PA for a week).

Exclusion Criteria:

* smokers.
* free from any metabolic diseases such as hypertension, dyslipidaemia, and hyperglycaemia.
* not using any medication or substance known to influence cardiorespiratory or metabolic responses to exercise
* previously participated in a specific training program within the past 6 months before the exercise interventions.
* contraindications to exercise based on the Physical Activity Readiness Questionnaire (PAR-Q) such as musculoskeletal injuries.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: Height | Baseline only (Session 1)
  Standing height will be measured using a stadiometer with participants barefoot and standing in the anatomical position. The value used for analysis will be the height recorded at baseline (Session 1).Unit of Measure: centimeters (cm)
Outcome Measure: Body Weight | Session 1 (Week 0), Session 15 (Week 5), Session 30 (Week 10)
  Body weight will be measured using a calibrated digital scale with participants wearing light clothing and no shoes. The value used for analysis will be the body weight recorded at baseline (Session 1).Unit of Measure: kilograms (kg)
Outcome Measure: Body Mass Index (BMI) | Session 1 (Week 0), Session 15 (Week 5), Session 30 (Week 10)
  BMI will be calculated using height and weight measured at baseline, using the formula BMI = weight (kg) / height (m²). The final reported value will be the BMI calculated at Session 1.Unit of Measure: kg/m²
Change in Affective Valence During Low-Volume High-Intensity Interval Exercise | Measured at every training session (Sessions 1-30) over 10 weeks; primary analysis compares Sessions 1, 15, and 30
  Affective valence is assessed using the Feeling Scale (range -5 to +5) during each low-volume high-intensity interval exercise (Lv-HIIE) session, which consists of 6-10 cycles of 60 s shuttle running and 75 s active recovery. Affective valence is measured 5 minutes before exercise, 20 seconds before the end of warm-up, immediately after each 60-second work interval, and after cool-down during Sessions 1, 15, and 30. The reported value will be the mean change in Feeling Scale score from Session 1 to Session 30, with Session 15 serving as a mid-intervention reference time point.Feeling Scale score (-5 to +5)
Change in Felt Arousal During Low-Volume High-Intensity Interval Exercise | Measured at every training session (Sessions 1-30) over 10 weeks; primary analysis compares Sessions 1, 15, and 30
  Felt arousal is assessed using the Felt Arousal Scale (range 1 to 6) during Lv-HIIE sessions (6-10 cycles of 60 s work + 75 s active recovery). Felt arousal is measured 5 minutes before exercise, 20 seconds before the end of warm-up, immediately after each 60-second work interval, and after cool-down during Sessions 1, 15, and 30. The reported value will be the mean change in Felt Arousal Scale score from Session 1 to Session 30, with Session 15 as a mid-intervention reference.Felt Arousal Scale score (1-6)
Change in Rating of Perceived Exertion During Low-Volume High-Intensity Interval Exercise | Measured at every training session (Sessions 1-30) over 10 weeks; primary analysis compares Sessions 1, 15, and 30
  Rating of perceived exertion (RPE) is measured using the Borg 6-20 scale during Lv-HIIE sessions (6-10 cycles of 60 s work + 75 s active recovery). RPE is recorded 5 minutes before exercise, 20 seconds before the end of warm-up, immediately after each 60-second work interval, and after cool-down during Sessions 1, 15, and 30. The reported value will be the mean change in RPE from Session 1 to Session 30, with Session 15 as a mid-intervention reference point.Borg RPE score (6-20)
Change in Perceived Recovery During Low-Volume High-Intensity Interval Exercise | Measured at every training session (Sessions 1-30) over 10 weeks; primary analysis compares Sessions 1, 15, and 30
  Perceived recovery is assessed using the Perceived Recovery Scale (range 0 to 10) during Lv-HIIE sessions. It is measured immediately after each 75-second active recovery interval in every cycle during Sessions 1, 15, and 30. The reported value will be the mean change in Perceived Recovery Scale score from Session 1 to Session 30, with Session 15 as a mid-intervention reference.Perceived Recovery Scale score (0-10)
Change in Exercise Enjoyment During Low-Volume High-Intensity Interval Exercise | Measured at the end of Sessions 1, 15, and 30 over 10 weeks
  Exercise enjoyment is assessed using a validated enjoyment scale (range 1 to 7) at the end of the Lv-HIIE session. Enjoyment is measured once at the end of Sessions 1, 15, and 30. The reported value will be the change in enjoyment score from Session 1 to Session 30, with Session 15 as a mid-intervention reference.Enjoyment scale score (total 126 scores)
Change in Heart Rate During Low-Volume High-Intensity Interval Exercise | Measured at every training session (Sessions 1-30) over 10 weeks; primary analysis compares Sessions 1, 15, and 30
  Heart rate is measured continuously and summarized at specific time points (5 minutes before exercise, 20 seconds before the end of warm-up, immediately after each 60-second work interval, and after cool-down) during Lv-HIIE sessions (6-10 cycles of 60 s work + 75 s active recovery). Heart rate is recorded during Sessions 1, 15, and 30. The reported value will be the mean change in heart rate (beats per minute) from Session 1 to Session 30, with Session 15 as a mid-intervention reference.Beats per minute (bpm)
Change in Heart Rate Recovery During Low-Volume High-Intensity Interval Exercise | Measured at every training session (Sessions 1-30) over 10 weeks; primary analysis compares Sessions 1, 15, and 30
  Heart rate recovery is assessed as heart rate measured immediately after each 75-second active recovery interval during Lv-HIIE sessions. Heart rate recovery is recorded for all cycles in Sessions 1, 15, and 30. The reported value will be the mean change in heart rate recovery (beats per minute during recovery periods) from Session 1 to Session 30, with Session 15 as a mid-intervention reference.Beats per minute (bpm)
Psychophysiological Stress (Blood Biomarkers) | Day 1 (Week 1, baseline), Day 15 (Week 5), and Day 30 (Week 10, final assessment), with samples collected pre-exercise, immediately post-exercise, and 30 minutes post-exercise
  Psychophysiological stress will be assessed using venous blood biomarkers. Blood samples will be collected at three predefined assessment days during the 10-week intervention: Day 1 (Week 1, baseline), Day 15 (Week 5), and Day 30 (Week 10, final assessment).
  At each assessment day, venous blood will be drawn at three standardized time points:
  Immediately before exercise (pre-exercise) Immediately after exercise (0 minutes post-exercise) 30 minutes post-exercise This results in nine total blood draws per participant. Biomarkers include cortisol, ACTH, and related stress markers. Changes will be compared across these assessment days.Concentration (pg/mL or ng/mL)
Goal Orientation in Exercise Measure (GOEM) Total Score | Baseline (Day 1, before the first training session)
  Goal orientation will be assessed using the Goal Orientation in Exercise Measure (GOEM), a validated 10-item questionnaire scored on a 5-point Likert scale (1-5). Item scores are summed to produce a total GOEM score ranging from 0 to 50. The questionnaire is completed once at baseline, before the first training session, to characterize individual differences in goal-orientation tendencies that may influence perceptual and physiological responses during the intervention. The reported value will be the total GOEM score.Score range 0-50
Connor-Davidson Resilience Scale (CDRS) Total Score | Baseline (Day 1, before the first training session)
  Psychological resilience will be assessed using the Connor-Davidson Resilience Scale (CDRS), a validated resilience questionnaire producing a total score ranging from 0 to 100. The scale is administered once at baseline, prior to the first training session, to evaluate individual differences in resilience traits that may influence perceptual and physiological responses during the intervention. The reported value will be the total CDRS score.Score range 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Sains Malaysia, Health Campus, Complex sports center, Kota Bharu, Kelantan, Malaysia